CLINICAL TRIAL: NCT01297621
Title: Satisfaction, Physical Activity and Sexuality Outcomes in Breast Reduction Patients
Brief Title: Physical Activity and Sexuality After Reduction Mammaplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniela Francescato Veiga (Other)
Responsible Party: Sponsor-Investigator, Daniela Francescato Veiga, Professor, Federal University of São Paulo
Organization: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Mestre 1; 0651/10 (Other: Ethical Commitee)
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Breast Hypertrophy
Keywords: breast hypertrophy; physical activity; sexuality; patient satisfaction
MeSH Terms: conditions — Gigantomastia; Motor Activity; Sexuality; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breast reduction (Experimental): Breast hypertrophy women allocated to this arm will undergo reduction mammaplasty
  Interventions: Procedure: reduction mammaplasty
- Control (Other): Patients in this arm will be assessed twice, without surgical intervention
  Interventions: Other: control

INTERVENTIONS:
Procedure: reduction mammaplasty — conventional reduction mammaplasty
  Arms: Breast reduction
Other: control — follow up, questionnaire responses
  Arms: Control

SUMMARY:
This prospective controlled trial was designed to determine whether breast reduction may influence physical activity and sexuality of breast hypertrophy women.

DETAILED DESCRIPTION:
Breast hypertrophy is a frequent condition among women; reduction mammaplasty is one of the most performed procedures in plastic surgery.Previous studies have demonstrated that breast hypertrophy is associated to back pain, and patients often complain about physical limitations due to this condition, as well as sexual impairment. Thus, this trial was designed to test the hypothesis that reduction mammaplasty may improve physical and sexual performance of breast hypertrophy patients,and patients'satisfaction with the results of the operation. Three validated tools were used: the International Physical Activity Questionnaire (IPAQ), the Female Sexual Quotient and the Breast Evaluation Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* breast hypertrophy
* candidate to reduction mammaplasty
* body mass index under 30Kg/m2
* women with sexual activity

Exclusion Criteria:

* pregnancy, delivery or breast feeding during the last 12 months
* body mass index over 30Kg/m2
* breast cancer history
* previous breast surgery
* smoking

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
physical activity | 6 months
  Physical activity will be assessed by a validated instrument, the International Physical Activity Questionnaire (IPAQ), at pre-operative and 6 months after breast reduction

SECONDARY OUTCOMES:
Patient's satisfaction | 6 months
  Patient's satisfaction will be assessed after 6 months, by the Breast Evaluation Questionnaire
Sexuality | 6 months
  Sexuality will be assessed by a brazilian validated questionnaire, the Female Sexual Quotient, at preoperative and sixth postoperative month

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa L Resende, MD, Principal Investigator — Federal University of São Paulo; Miguel Sabino-Neto, MD, PhD, Study Director — Federal University of São Paulo; Daniela F Veiga, MD, PhD, Study Director — Federal University of São Paulo; Lydia M Ferreira, MD, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Hospital São Paulo, São Paulo, São Paulo, Brazil